CLINICAL TRIAL: NCT04593485
Title: Single-center, Open-label, Single-arm Phase II Clinical Trial of Anti-PD-1 Antibody (Camrelizumab for Injection) in the Treatment of Patients With Malignant Melanoma of the Female Genital Tract
Brief Title: Anti-PD-1 Antibody in the Treatment of Patients With Malignant Melanoma of the Female Genital Tract
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-GYN-006
Record Dates: First submitted 2020-08-18; First posted 2020-10-20 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — camrelizumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): patients with postoperative recurrence of malignant melanoma of the female genital tract requiring adjuvant therapy, Camrelizumab for injection
  Interventions: Drug: Camrelizumab for injection
- Cohort 2 (Experimental): patients with metastatic or unresectable malignant melanoma of the female genital tract, Camrelizumab for injection
  Interventions: Drug: Camrelizumab for injection

INTERVENTIONS:
Drug: Camrelizumab for injection — Carrelizumab will be administered at a fixed dose
  Other Names: Jiangsu Hengrui, SHR-1210

SUMMARY:
This is a single-center, open-label, single-arm phase II clinical study to exploratory observe and evaluate the efficacy and safety of anti-PD-1 antibody (Camrelizumab for Injection) in patients with malignant melanoma of the female genital tract.

Subjects were to have a safety visit 3 days prior to dosing in each treatment cycle after the study. Imaging was performed every 8 weeks to assess efficacy until radiographic progression, initiation of new antineoplastic therapy, withdrawal of consent, or subject lost to follow-up/death.

After the end of treatment, an end-of-treatment visit and a post-treatment safety visit will also be performed. After the end of treatment, subjects will also be followed up for survival (every 3 months for years 1 to 2, every 4 months for years 3, every 6 months for years 4 to 5, and annually from year 6) to collect and record the survival status of subjects and subsequent anti-tumor treatment.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm phase II clinical study to exploratory observe and evaluate the efficacy and safety of anti-PD-1 antibody (Camrelizumab for Injection) in patients with malignant melanoma of the female genital tract.

The patients were divided into two cohorts according to their conditions: Cohort 1: patients with postoperative recurrence of malignant melanoma of the female genital tract requiring adjuvant therapy；Cohort 2: patients with metastatic or unresectable malignant melanoma of the female genital tract who were screened eligible and received study treatment after being fully informed and signing the informed consent form.

Camrelizumab will be administered at a fixed dose of 200 mg intravenously (iv) on D1 in a 14-day cycle. All subjects will be administered until they reach the end of treatment standard specified in the protocol.

Subjects were to have a safety visit 3 days prior to dosing in each treatment cycle after the study. Imaging was performed every 8 weeks to assess efficacy until radiographic progression, initiation of new antineoplastic therapy, withdrawal of consent, or subject lost to follow-up/death.

After the end of treatment, an end-of-treatment visit and a post-treatment safety visit will also be performed. Subjects who have concluded the study treatment for reasons other than disease progression will receive imaging assessment at the end of treatment (if imaging evaluation is not performed at 4 months) and imaging assessment every 3 months after the end of treatment to assess the time to disease progression. After the end of treatment, subjects will also be followed up for survival (every 3 months for years 1 to 2, every 4 months for years 3, every 6 months for years 4 to 5, and annually from year 6) to collect and record the survival status of subjects and subsequent anti-tumor treatment.

Tumor tissue samples, sections, paraffin blocks or biopsy blocks, and biomarkers, including but not limited to PD-L1 expression level and the proportion of positive cells, TMB level and MMR status, will be collected from subjects during the screening period after the most recent previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join this study and sign the informed consent form;
* Age: women aged 18 to 70 years;
* Cohort 1 patients need to meet: radical surgery in our hospital or other hospital, no gross residual lesions or imaging metastases; and our hospital surgical histopathology (or pathology consultation in our hospital) confirmed as patients with primary genital tract melanoma (vulva, vagina, cervix or uterine body origin); for vulvar malignant melanoma: postoperative pathology suggests tumor breslow thickness ≥ 1.5 mm or lymph node metastasis, in line with any of the above can be enrolled; for vaginal malignant melanoma: postoperative pathology suggests tumor diameter > 3 cm, depth of invasion ≥ 1/2 or tumor breslow thickness ≥ 2 mm, lymph node metastasis, in line with any of the above can be enrolled; for cervical or uterine body malignant melanoma: all patients after radical surgery can be enrolled. Cohort 2 patients should meet: patients with primary female genital tract melanoma confirmed by histopathology (or pathology consultation in our hospital), who are recurrent metastatic disease or unresectable after initial treatment, and have at least one measurable lesion (RECIST version 1.1);
* If the investigator considers that the scope of surgery is too large, patients can be considered for neoadjuvant anti-PD-1 antibody therapy (no more than 4 cycles) + interval surgery + postoperative adjuvant anti-PD-1 antibody therapy: patients receiving neoadjuvant therapy must receive interval surgery after 3-4 cycles of treatment. Confirmation of pathological diagnosis using mandatory biopsy tissue samples (e.g. obtained by hollow core needle, biopsy, excision, etc.);
* 5-10 formalin-fixed, paraffin-embedded tumor tissue sections from lesions that can be obtained (not required) for biomarker analysis;
* ECOG-PS score: 0-1;
* Expected survival time ≥ 12 weeks;
* Bone marrow function: neutrophils ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90 g/L;
* Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal; AST and ALT ≤ 2.5 times the upper limit of normal or the presence of liver metastasis ≤ 5 times the upper limit of normal; total bilirubin ≤ 1.5 times the upper limit of normal, or patients with Gilbert's syndrome ≤ 2.5 times the upper limit of normal;
* Non-surgically sterilized subjects of childbearing age must agree to take effective contraceptive measures during the study treatment and within 3 months after the end of the study treatment period; Non-surgically sterilized women of childbearing age must have a negative serum or urine pregnancy test before the study;
* Non-lactating patients.

Exclusion Criteria:

* Patients with central nervous system disease or brain metastases; patients who have received systemic, radical treatment of brain or meningeal metastases (radiotherapy or surgery), such as imaging confirmed stable has been maintained for at least 1 month, and have stopped systemic hormone therapy (dose > 10 mg/day prednisone or other effective hormones) for more than 2 weeks, no clinical symptoms can be included;
* Other malignant tumors occurred in the past 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer;
* The researchers believe that will affect the ability of subjects to receive the study program treatment, and uncontrolled serious medical diseases, such as severe medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension (after treatment: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, Based on the average of BP readings obtained by ≥ 2 measurements), uncontrolled infection, active peptic ulcer, etc.;
* Known interstitial lung disease or history or evidence of non-infectious pneumonia treated with corticosteroids; or patients who may interfere with the detection or treatment of suspected drug-related pulmonary toxicity;
* Known allergy, high sensitivity or intolerance to study-related drugs or their excipients;
* received other experimental drugs or participated in other clinical studies for the purpose of anti-cancer therapy within 30 days before the first dose;
* Serious infection occurred before the start of study treatment, including but not limited to infectious complications requiring hospitalization, bacteremia or severe pneumonia;
* Previously received anti-programmed cell death-1 (PD-1), anti-PD-L1, anti-CD137 or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody therapy;
* 7 days before receiving the study drug, diagnosed with immunodeficiency disease or receiving systemic steroid therapy or other immunosuppressive therapy;
* patients with active pulmonary tuberculosis;
* syphilis patients;
* human immunodeficiency virus (HIV) positive;
* hepatitis B surface antigen positive (HBsAg), and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV-DNA) test ≥ 1 × 103 IU/mL subjects; if HBsAg positive, and peripheral blood HBV-DNA < 1 × 103 IU/mL, if the investigator believes that the subject is in a stable period of chronic hepatitis B and will not increase the risk of subjects, Subjects are eligible;
* Hepatitis C virus (HCV) antibody positive and HCV RNA test positive.
* less than 4 years before the study medication or may be vaccinated during the study;
* the researchers determine that patients who are not suitable for this study, such as alcoholism, drug abuse, other serious diseases (including mental illness) need combined treatment, there are serious laboratory abnormalities, accompanied by family or social factors, will affect the safety of patients or data and sample collection;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | RFS was defined as the time from surgery to first local, regional, or distant tumor recurrence or death from any cause, whichever came first, assessed up to one year.
  The primary endpoint for Cohort 1 is relapse-free survival (RFS)
Objective Response Rate (ORR) | Tthrough study completion, an average of 2 year.
  The primary endpoint for Cohort 2 is Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Adverse events (AEs) | Through study completion, an average of 2 year.
  according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Principal Investigator — Fudan University Shanghai Cancer Centre
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai